CLINICAL TRIAL: NCT00679029
Title: Adjuvant Doxorubicin, Cyclophosphamide Followed by Avastin Given With Paclitaxel and Gemcitabine for Stage II and III Breast Cancer That Does Not Over-express Human Epidermal Growth Factor Receptor 2 (HER-2)/Neu
Brief Title: Chemotherapy & Bevacizumab for Human Epidermal Growth Factor Receptor 2 (HER2)/Neu-Negative Stage II/III Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: drug toxicity
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0412-07-FB; NCI-2009-01693 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA036727 (NIH)
Record Dates: First submitted 2008-05-15; First posted 2008-05-16 (Estimated); Results first posted 2018-12-12 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: HER2-negative Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Doxorubicin; Cyclophosphamide; Bevacizumab; Paclitaxel; Taxes; Gemcitabine; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemotherapy with Bevacizumab (Experimental): Doxorubicin 60 mg /M2 followed by cyclophosphamide 600 mg/M2 (AC) will be given every 2 weeks for cycles 1-4.
  Paclitaxel 175 mg/M2 followed by gemcitabine 1500 mg/M2 (TG) will be given every 2 weeks for cycles 5-8.
  Beginning cycle 5, B1= Avastin 10 mg/kg will be given as a single IV dose following each TG treatment every 2 weeks for cycles 5-7.
  Interventions: Drug: doxorubicin hydrochloride; Drug: cyclophosphamide; Biological: bevacizumab; Drug: paclitaxel; Drug: gemcitabine hydrochloride; Other: laboratory biomarker analysis; Biological: pegfilgrastim

INTERVENTIONS:
Drug: doxorubicin hydrochloride — Given IV
  Other Names: ADM; ADR; Adria; Adriamycin PFS; Adriamycin RDF
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
Drug: paclitaxel — Given IV
  Other Names: Anzatax; Asotax; TAX; Taxol
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar
Other: laboratory biomarker analysis — Correlative studies
Biological: pegfilgrastim — Given subcutaneously
  Other Names: Filgrastim SD-01; GCSF-SD01; Neulasta; SD-01 sustained duration G-CSF

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as doxorubicin hydrochloride, cyclophosphamide, paclitaxel, and gemcitabine hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of breast cancer by blocking blood flow to the tumor. Giving combination chemotherapy together with bevacizumab after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase II trial is studying the side effects and how well giving combination chemotherapy together with bevacizumab works in treating women with HER2/neu-negative stage II or stage III breast cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the feasibility of administering two sequential chemotherapy doublets with Avastin in the adjuvant setting.

II. To assess the safety of Avastin in the adjuvant setting particularly regarding cardiac function, wound healing and toxicity of radiation.

SECONDARY OBJECTIVES:

I. To determine the effect of Avastin on immunity, especially Vascular endothelial growth factor A (VEGF-A) upregulation of myeloid-derived suppressor cells (MDSC) and suppression of T-Cells.

II. To determine the effect of therapy on numbers of myeloid derived suppressor cells and compare the humoral and cellular response to p53 in breast cancer patients treated with the same chemotherapy.

III. Patients will be followed for freedom from tumor progression and survival.

OUTLINE:

COURSES 1-4: Patients receive doxorubicin hydrochloride IV and cyclophosphamide IV on day 1 and pegfilgrastim subcutaneously (SC) on day 1. Treatment repeats every 2 weeks for 4 courses in the absence of unacceptable toxicity or disease progression.

COURSES 5-7: Patients receive paclitaxel IV and gemcitabine hydrochloride IV on day 1 and pegfilgrastim SC on day 1. Patients also receive bevacizumab IV on day 1 in courses 5-7. Treatment repeats every 2 weeks for 4 courses in the absence of unacceptable toxicity or disease progression.

COURSES 8-16: Patients receive bevacizumab IV alone on day 1. Treatment repeats every 3 weeks for 8 courses in the absence of unacceptable toxicity or disease progression.

After course 8, patients may undergo radiotherapy and hormone therapy, if clinically indicated.

After completion of study treatment, patients are followed every 3 months for 2 years and then every 6 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of invasive breast cancer: By pathologic evaluation, primary tumor must be T1-4N1-3M0 or T3-4N 0M0 that is ER/PR positive or negative and HER-2/neu negative (1+) immunocytochemistry or not amplified by Fluorescence in situ hybridization (FISH)
* OR By pathologic evaluation, primary tumor must be T2N0 that is estrogen receptor (ER), progesterone receptor (PR) and HER-2neu negative
* Women of reproductive potential must be non-pregnant and non-nursing and must agree to employ an effective barrier method of birth control throughout the study and for up to 6 months following treatment
* Women of child-bearing potential, must have a negative pregnancy test within 7 days of initiating study (no childbearing potential is defined as age 55 years or older and no menses for two years or any age with surgical removal of the uterus and/or both ovaries)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Definitive surgery, lumpectomy and axillary sampling or modified radical mastectomy
* Three weeks since last surgery other than port or right atrial catheter placement
* No significant cardiac disease and a normal left ventricular ejection fraction
* No significant open wounds, uncontrolled hypertension, history of venous or arterial clotting
* Adequate laboratory parameters within 30 days prior to enrollment defined as:
* Absolute neutrophil count greater than or equal to 1,500/mcl
* Platelet count equal to or greater than 150,000/mcl
* Hemoglobin >11gm/dl
* Alkaline phosphatase equal or less than 1.5 times the upper limit normal (ULN)
* Total bilirubin equal to or less than 1.5 times the ULN
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) no greater than 1.5 times the ULN
* Creatinine less than 1.5 times the ULN
* Urine protein < 2+ on urinalysis, UPC 1.0 or 24 hour urine < 1 g protein
* No active serious infections or other condition precluding chemotherapy
* Able to give informed consent
* Able to return for treatment and follow-up on the specified days

Exclusion Criteria:

* Prior malignancy; except for adequately treated basal cell or squamous cell skin cancer or noninvasive carcinomas, or other cancer from which the patient has been disease free for 5 years
* Prior chemotherapy or radiation therapy
* Breast cancer that over expresses Her-2/neu
* Stage IV or metastatic breast cancer
* Inability to cooperate with treatment protocol
* Any comorbidity or condition which, in the opinion of the investigator, may interfere with the assessments and procedures of this protocol
* Inadequately controlled hypertension (defined as systolic blood pressure > 150 and/or diastolic blood pressure > 100 mmHg on antihypertensive medications
* Any prior history of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* History of myocardial infarction or unstable angina within 12 months of study enrollment
* Any history of stroke or transient ischemic attack at any time
* Significant vascular disease (e.g., aortic aneurysm, aortic dissection)
* Symptomatic peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study enrollment
* Serious, non-healing wound, ulcer, or bone fracture
* Proteinuria at screening as demonstrated by either urine protein/creatinine (UPC) ratio >= 1.0 at screening OR urinalysis for proteinuria >= 2+ (patients discovered to have >= 2+ proteinuria on urinalysis at baseline and undergo a 24 hour urine collection and demonstrate > 1g of protein in 24 hours are ineligible)
* Known hypersensitivity to any component of Avastin or gemcitabine or other required drugs in the study
* History of venous or arterial thrombosis
* Current, ongoing treatment with full-dose warfarin or its equivalent (i.e., unfractionated and/or low molecular weight heparin) for any reason (ASA okay)

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-05-02 (Actual); Primary Completion 2010-11-18 (Actual); Study Completion 2010-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth C Reed, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemotherapy With Bevacizumab: Doxorubicin 60 mg /M2 followed by cyclophosphamide 600 mg/M2 (AC) will be given every 2 weeks for cycles 1-4.
  Paclitaxel 175 mg/M2 followed by gemcitabine 1500 mg/M2 (TG) will be given every 2 weeks for cycles 5-8.
  Beginning cycle 5, B1= Avastin 10 mg/kg will be given as a single IV dose following each TG treatment every 2 weeks for cycles 5-7.
  N=Growth factor pegfilgrastim 6 mg will be administered subcutaneously on day 1 after AC and TG treatment every 2 weeks for 8 cycles.
Period: Overall Study
Arm/Group | Chemotherapy With Bevacizumab
Started | 15
Completed | 10
Not Completed | 5
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm I: AC = Doxorubicin 60 mg /M2 followed by cyclophosphamide 600 mg/M2 will be given every 2 weeks for cycles 1-4.
  TG = Paclitaxel 175 mg/M2 followed by gemcitabine 1500 mg/M2 will be given every 2 weeks for cycles 5-8.
  Beginning cycle 5, B1= Avastin 10 mg/kg will be given as a single IV dose following each TG treatment every 2 weeks for cycles 5-7.
  N=Growth factor pegfilgrastim 6 mg will be administered subcutaneously on day 1 after AC and TG treatment every 2 weeks for 8 cycles.
Arm/Group | Arm I
Number analyzed (Participants) | 15
Age, Customized [Count of Participants; unit: Participants]
  >=19 years of age | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 12
  Black, Not Hispanic | 3
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Study Drug-associated Adverse Events Leading to Dose Holds or Reductions
Description: This outcome is to measure the feasibility of the of administering two sequential chemotherapy doublets with Avastin in the adjuvant setting in women with stage II and III breast cancer that does not over-express human epidermal growth factor receptor 2 (HER 2)/neu
Time Frame: through study completion, an average of 10 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I
Number analyzed (Participants) | 15
percentage of participants | 20 [4.33 to 48.09]

2. Primary Outcome: Count of Participants With Related Serious Adverse Events (SAEs) by NCI Common Toxicity Criteria v3.0
Description: Assess the safety of Avastin in the adjuvant setting particularly regarding cardiac function, wound healing and toxicity of radiation.
Time Frame: through study completion, an average of 10 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 15
Participants | 0

3. Secondary Outcome: Overall Survival as Assessed by the Kaplan and Meier Method
Description: Overall survival as assessed by the Kaplan and Meier method at 5 years
Time Frame: Original time frame: Up to 5 years from date of first treatment; study terminated at 2.5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I
Number analyzed (Participants) | 15
percentage of participants | 69.1 [36.7 to 87.3]

4. Secondary Outcome: Disease-free Survival
Description: Disease-free survival as assessed by the Kaplan and Meier method
Time Frame: From the date of first treatment to the date of disease progression/recurrence, second cancer, or death, whichever came first: Original time frame up to 5 years from date of first treatment; study terminated at 2.5 years
Population: estimated disease free survival at 5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I
Number analyzed (Participants) | 15
percentage of participants | 70 [38.2 to 87.6]

ADVERSE EVENTS:
Time Frame: Adverse events were collected during Avastin treatment, during a post-treatment follow-up period (approximately 30 weeks) and survival (original time frame: Up to 5 years from date of first treatment; study terminated at 2.5 years)
Arm/Group | Arm I
All-Cause Mortality (participants affected / at risk) | 1/15
Serious Adverse Events (participants affected / at risk) | 4/15
Other Adverse Events (participants affected / at risk) | 13/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=15)
colonic perforation (Gastrointestinal disorders) | 1 (1)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung Infection (Infections and infestations) | 1 (1) — pneumonia
Other, Weakness (General disorders) | 1 (1)
Other, alveolar hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Platelet count decrease (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Other, enteritis (Gastrointestinal disorders) | 1 (1)
Other, cellulitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=15)
Anemia (Blood and lymphatic system disorders) | 3 (6)
dermatitis radiation (Injury, poisoning and procedural complications) | 3 (3)
hyperglycemia (Metabolism and nutrition disorders) | 3 (3)
diarrhea (Gastrointestinal disorders) | 2 (2)
mucositis oral (Gastrointestinal disorders) | 2 (2)
proteinuria (Renal and urinary disorders) | 1 (1)
hypertension (Vascular disorders) | 3 (3)
weight gain (Investigations) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 (2)
White blood cell decreased (Investigations) | 3 (5)
neutrophil count decreased (Investigations) | 3 (5)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
fatigue (General disorders) | 2 (2)
myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Other - respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
platelet count decreased (Investigations) | 2 (5)
hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2)
hypoalbuminia (Metabolism and nutrition disorders) | 1 (2)
dehydration (Metabolism and nutrition disorders) | 1 (1)
Other - cellulitis (Musculoskeletal and connective tissue disorders) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes